CLINICAL TRIAL: NCT00987168
Title: Replace Sandostatine® in Three Daily Subcutaneous Injections by a Single Intramuscular Injection of Sandostatine® LP Per Month in Patients With a Diffuse Form of Hyperinsulinism
Brief Title: Sandostatine® LP and Hyperinsulinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC 07024
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2010-10

CONDITIONS: Congenital Hyperinsulinism
Keywords: Congenital Hyperinsulinism; Hypoglycemia,; Sandostatine subcutaneous in 3 daily injections; Intramuscular injection of Sandostatine® LP per month
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sandostatine LP (Experimental)
  Interventions: Drug: Sandostatine LP

INTERVENTIONS:
Drug: Sandostatine LP — Intramuscular injection of Sandostatine LP, once per month Dosage : 10 mg, 20 mg, 30 mg

SUMMARY:
To replace Sandostatine® in three daily subcutaneous injections by a single intramuscular injection of Sandostatine® LP per month in patients with a diffuse form of hyperinsulinism.

DETAILED DESCRIPTION:
Persistent hyperinsulinemic hypoglycemias of infancy (HI) are characterized by an inappropriate secretion of insulin responsible for profound hypoglycemias which require aggressive treatment to prevent severe and irreversible brain damage.

Thanks to the complementarity and to the synergy between paediatricians, paediatric surgeons, radiologists, pathologists and geneticists, an important stage was reached: the recognition of two clinically similar forms of HI but requiring a radically different treatment: a diffuse form and a focal form in the pancreas.

The medical treatment is based on proglycem, or diazoxide, then octreotide (Sandostatine ®, Novartis) with a dose of 10 to 50 µg/Kg/jour divided to three subcutaneous injections. Most neonates are resistant to diazoxide and side effects are observed (important edema and hypertrichosis). The Sandostatine® is a much more effective treatment, unfortunately with a short half-life and painful injections. In the cases of resistance to the medical treatment, the distinction of the two forms is essential to guide the surgical treatment : partial pancreatectomy in the focal forms, curing definitively hypoglycemia; subtotal pancreatectomy in the diffuse forms resisting to the medical treatment, leading to a diabetes and a pancreatic exocrine insufficiency. Also, the medical treatment is essential in the case of the diffuse forms to avoid a subtotal pancreatectomy. Mutations in two genes encoding the potassium channels, SUR1 and KIR6.2, are responsible for hyperinsulinism resistant to diazoxide.

The Sandostatine® marketed by Novartis exists in two forms, a "rapid" form and a "retarded liberation form". These two molecules have been approved in the treatment of adults in the following indications:

* Treatment of the clinical symptoms of digestive endocrine tumours
* Treatment of acromegaly
* Treatment of primitive thyrotrope adenomata
* Treatment of unfunctional adenoma
* Treatment of corticotrope adenoma during (Nelson syndrome) and of functional gonadotrope adenomata
* After pancreatic surgery
* Emergency treatment of bleeding secondary to cirrhosis.

Sandostatine® has neither approval for hyperinsulinism, nor in children even though many international publications reported efficacy of treatment by Sandostatine® in hyperinsulinemic children since 1983. Also, by consensus most international teams taking care of hyperinsulinism in infancy propose this treatment to their patients.

Ten children who have a diffuse form of hyperinsulinism have been treated in our department by Sandostatine® given in three subcutaneous injections for several years, in order to avoid a sub-total pancreatectomy. The only possible adverse effect is the appearance of vesicular lithiasis which can be treated by ursodesoxycholic acid . We changed the Sandostatine® treatment of one of our patients by the Sandostatine® LP (retarded liberation form) after written consent of his two parents. Thus we could stop the three injections per day of Sandostatine®. Sandostatine® LP proved to be as efficient on hypoglycemias as the subcutaneous multi-daily injections (SC). The glycemia values were strictly normal, and no hypoglycaemia was observed. Following this observation, we propose to try to substitute the treatment of Sandostatine® given in several subcutaneous injections by one injection of Sandostatine® LP in 10 children followed in the department of Metabolism for hyperinsulinism.

The awaited result of this study is to demonstrate efficacy of Sandostatine® LP and thus replace Sandostatine® in three daily subcutaneous injections by a single intramuscular injection of Sandostatine® LP per month. This study will contribute to an undeniable improvement of the quality of life for the patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* congenital hyperinsulinism patients
* age of patients : 6 months to 16 years
* normoglycemia under sandostatine subcutaneous
* contraception efficiency
* signed informed consent

Exclusion Criteria:

* refusal from parents
* vesicular lithiasis
* absence of social security
* hypersensitivity to octreotide or excipients
* pregnancy or nursing mother

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Glycemia > or equal to 3 mmol/L, before and after 4 meals +Midnight + 4 am | 6 months

SECONDARY OUTCOMES:
Abdominal ultra echography, before and after 6 month treatment | 6 months
Life quality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascale De Lonlay, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker Hospital, Paris, France